CLINICAL TRIAL: NCT07021300
Title: Early Versus Interval Laparoscopic Cholecystectomy for Acute Cholecystitis
Acronym: EILC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr. Waseem Ullah, Registrar, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ref: No. 863/LRH/ MTI; 863/LRH/MTI (Other: Lady Reading Hospital Ethical Review Committee)
Record Dates: First submitted 2025-05-30; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Acute Cholecystitis; Cholelithiasis; Gallbladder Diseases
Keywords: Randomized controlled trial; Laparoscopic cholecystectomy; Acute cholecystitis; Early surgery; Delayed surgery
MeSH Terms: conditions — Cholecystitis, Acute; Cholelithiasis; Gallbladder Diseases

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: early laparoscopic cholecystectomy (within 72 hours) or interval laparoscopic cholecystectomy (after 4 weeks).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors collecting data on operative time, hospital stay, and conversion rates were blinded to group allocation. Complete blinding of participants and surgeons was not feasible due to the nature of the surgical timing intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Laparoscopic Cholecystectomy (Experimental): Patients in this arm will undergo laparoscopic cholecystectomy within 72 hours of diagnosis of acute cholecystitis. Surgery will be performed using a standard four-port technique under general anesthesia by an experienced surgeon.
  Interventions: Procedure: Early Laparoscopic Cholecystectomy
- Interval Laparoscopic Cholecystectomy (Active Comparator): Patients in this arm will receive initial conservative management, including antibiotics and analgesics, followed by laparoscopic cholecystectomy performed after 4 weeks. The surgery will also follow the standard four-port technique under general anesthesia.
  Interventions: Procedure: Interval Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Early Laparoscopic Cholecystectomy — A standard four-port laparoscopic cholecystectomy performed within 72 hours of diagnosis of acute cholecystitis. Surgery is done under general anesthesia by an experienced surgeon. This group receives no prolonged preoperative conservative management. Timing aligns with Tokyo Guidelines 2013 recommendation for early intervention
  Other Names: Early LC
  Arms: Early Laparoscopic Cholecystectomy
Procedure: Interval Laparoscopic Cholecystectomy — A standard four-port laparoscopic cholecystectomy performed after 4 weeks of initial conservative management with antibiotics and analgesics. The procedure is conducted under general anesthesia by the same experienced surgeon, using the same technique as the early group. This approach represents delayed surgical management per traditional protocols.
  Other Names: Interval LC
  Arms: Interval Laparoscopic Cholecystectomy

SUMMARY:
This study compares two different timing approaches for gallbladder removal surgery in patients with acute gallbladder inflammation (acute cholecystitis).

When someone develops acute cholecystitis, doctors need to remove the gallbladder using a minimally invasive technique called laparoscopic surgery. However, there is ongoing debate about the best timing for this surgery. Some doctors prefer to operate early (within 3 days of diagnosis), while others prefer to wait and operate later (after 4 weeks of medical treatment).

In this study, we randomly assigned 166 patients with acute cholecystitis to receive either:

* Early surgery: Laparoscopic gallbladder removal within 72 hours of diagnosis
* Delayed surgery: Laparoscopic gallbladder removal after 4 weeks of antibiotic treatment

All surgeries were performed by the same experienced surgeon using standard techniques. We measured how long each surgery took, how many days patients stayed in the hospital, and how often the surgeon needed to switch from the minimally invasive approach to open surgery.

The study found that patients who had early surgery had shorter operation times, went home from the hospital sooner, and were less likely to need open surgery compared to patients who waited 4 weeks for their operation.

This research helps doctors and patients make better decisions about the timing of gallbladder surgery when someone has acute cholecystitis.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to address the clinical question of optimal timing for laparoscopic cholecystectomy in acute cholecystitis, a condition affecting thousands of patients annually worldwide. The study was conducted in response to conflicting evidence and varying clinical practices regarding surgical timing.

Study Design and Setting:

The trial employed a parallel-group, single-blind randomized controlled design conducted at the General Surgery Department of Lady Reading Hospital, a tertiary care teaching hospital in Pakistan. The study period extended from May 1, 2024, to December 31, 2024, with comprehensive follow-up until patient discharge.

**Randomization and Blinding:** Participants were allocated using blocked randomization to ensure equal group sizes throughout the recruitment period. While complete blinding was not feasible due to the nature of the intervention, outcome assessors were blinded to group allocation during data collection. A computer-generated randomization sequence was used, with allocation concealment maintained through sealed opaque envelopes.

Intervention Protocols:

Group A (Early LC) patients underwent laparoscopic cholecystectomy within 72 hours of acute cholecystitis diagnosis. These patients were admitted, prepared for surgery with standard pre-operative protocols, and underwent surgery during the acute inflammatory phase.

Group B (Interval LC) patients received initial conservative management with intravenous antibiotics, analgesics, and supportive care during their index admission. After clinical improvement and discharge, they returned after 4 weeks for elective laparoscopic cholecystectomy during the quiescent phase.

Surgical Technique:

All procedures followed standardized protocols using the critical view of safety technique. The four-port approach included an umbilical port for the camera, a subxiphoid port for retraction, and two ports below the right costal margin for dissection and clipping. Calot's triangle dissection followed established principles with careful identification of the hepatocystic artery and cystic artery before clipping and division.

Outcome Measurement:

Primary outcomes were measured using standardized protocols. Operative time was recorded from anesthesia induction to complete abdominal wall closure using calibrated stopwatches. Hospital stay was calculated from surgery completion to consultant discharge decision. Conversion to open surgery was documented when the surgeon determined laparoscopic completion was unsafe or technically impossible.

**Quality Assurance:** A dedicated research fellow was assigned to each case for real-time data collection, ensuring accuracy and completeness. All procedures were performed by a single consultant surgeon with over five years of laparoscopic experience, eliminating surgeon-related variability. Post-operative care followed standardized protocols with daily assessments by the surgical team.

Statistical Considerations:

Sample size calculation was based on anticipated conversion rates from previous literature, with 80% power to detect a clinically meaningful difference. Effect modification analysis was pre-planned for key demographic and clinical variables to identify potential subgroup effects.

The study protocol received institutional review board approval and was conducted in accordance with Declaration of Helsinki principles, with comprehensive informed consent obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 60 years
* Diagnosis of acute cholecystitis confirmed by history (right hypochondrial pain <5 days), clinical examination (tenderness in right hypochondrium), and ultrasound (thickened fibrosed gallbladder wall)
* Presentation within 24 hours of symptom onset
* ASA physical status class I or II
* Provided written informed consent

Exclusion Criteria:

* Patients with stones in the common bile duct on ultrasound
* Patients with empyema of the gallbladder on ultrasound
* Severe comorbidities (e.g., uncontrolled diabetes, ASA class III or higher)
* Pregnancy
* Previous upper abdominal surgery
* Refusal to participate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intraoperatively (from anesthesia induction to closure of abdominal wall, assessed once during the surgery)
  Operative time measured in minutes from anesthesia induction to complete closure of the abdominal wall, recorded using a standardized stopwatch protocol.

SECONDARY OUTCOMES:
Length of Hospital Stay | Postoperatively (from end of surgery to discharge, assessed once at discharge)
  Postoperative hospital stay measured in full days from the time of surgery until the consultant surgeon's discharge decision.
Conversion to Open Surgery | Intraoperatively (assessed during the surgical procedure)
  Proportion of laparoscopic cholecystectomy cases that were converted to open cholecystectomy, as determined intraoperatively by the operating surgeon.

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study was not designed with data sharing agreements or participant consent for secondary data use. Ethical and institutional restrictions prevent public data release.